CLINICAL TRIAL: NCT04645771
Title: Safety and Efficacy Study of Endovenous Microwave Ablation for Treatment of Varicose Veins
Acronym: EMINENCE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Chunshui He, Director of Vascular Surgery in ChengduUTCM, Chengdu University of Traditional Chinese Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ChengduUTCMvs
Record Dates: First submitted 2020-10-31; First posted 2020-11-27 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Vascular Diseases, Peripheral; Venous Insufficiency of Leg; Varicose Veins of Lower Limb
Keywords: microwave ablation; varicose veins; traditional treatment
MeSH Terms: conditions — Peripheral Vascular Diseases; Varicose Veins | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: A total of 50 patients with varicose veins of lower extremities treated with microwave ablation catheter were selected to observe their venous closure rate and postoperative adverse reactions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Microwave ablations (Experimental): A total of 50 patients with varicose veins of lower extremities treated with microwave ablation catheter were selected to observe their annual venous closure rate and postoperative adverse reactions.
  Interventions: Procedure: Questionnaires

INTERVENTIONS:
Procedure: Questionnaires — Questionnaires to assess the quality of life (EQ-5D, CVVQ, CIVIQ, AVVQ, Patient satisfaction survey)

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of microwave ablation catheter in the treatment of varicose veins in lower extremities,meanwhile, to compare the quality of subjects'lives before and after treatment.

DETAILED DESCRIPTION:
The chronic venous insufficiency of lower extremities (chronic venous insufficiency, CVI) is a set of a series of clinical syndrome caused by venous reflux, common symptoms are heaviness, fatigue, swelling, burning sentation, itching, pain, etc.The main causes of superficial varicose veins are weakness of superficial vein wall, insufficiency or defect of vein valve closure and increased pressure inside veins.The weakness of venous wall, the decreasing of flexibility, venous valve defects the the poor structure, be related with genetic factor, belong to "primary" inferior venous valves' incomplete closure.The influencing factors of primary valve insufficiency include heavy physical labor, long standing or sitting work, obesity, pregnancy, chronic constipation, and chronic cough.Varicose veins secondary to a history of venous thrombosis of the lower extremities, venous system obstruction and increased venous pressure caused by circulating blood volume exceeding reflux load are secondary.When the valve of the great saphenous vein at the junction of the saphenous vein is damaged and closed incompletely, the valve function of the distal and perforating vein can be affected step by step, and the small saphenous vein can also be affected through its branch vein.Because the superficial vein wall's muscle layer is thin and their surrounding lackness of connective tissue, blood regurgitation can cause the venous lumen to thicken, tortuosity and lengthen, presenting as superficial varicose veins.Because of the severe venous pressure of lower extremity,the vascular permeability of football boots is increasing,resulting the appearance of a large number of blood capillary hyperplasia.Due to a large number of fibrinogen hindered the exchange between capillary and the surrounding tissue, the nutritional change of subcutaneous tissue occured,including skin pigmentation, eczema, dermatitis, subcutaneous lipid sclerosis and ulceration.

The traditional treatments of lower extremity varicose veins,including high ligation and stripping of great saphenous vein,varicose vein's resection and ligation of perforating vein,can cause large trauma,huge pain,limitation of activity and long convalescence and aesthetic problems,etc.As a consequence,a variety of minimally invasive method with small wound,little pain and early recovery are prevalently applied in clinical, also achieved plenty of good therapeutic effect.According to the different mechanism of minimally invasive treatment, it can be divided into two categories: physical injury (laser closure, radiofrequency closure, microwave treatment, electrocoagulation, transparent direct rotation, laparoscopic great saphenous vein resection, etc.) and chemical injury (sclerosing agent injection).

Clinical observation in our department found that the pain, bruising, numbness, and number of incisions after microwave ablation were all lower than those of traditional high position ligation and extraction with laser closure.

The purpose of this study is to report a monocentricity, prospective Chinese experience using the ECO Varicose Veins Therapeutic Unit from ECO (Nanjing ECO Microwave System Co.Ltd) for Endovenous Microwave Ablation (EMA) to treat primary great and short saphenous vein reflux and to evaluate its safety, efficacy and life quality.

ELIGIBILITY:
Inclusion Criteria:

- Age >18 years, and <90 years ,and able to understand the requirements of the study and provide informed consent and accept the exams and follow-up.

C2 - C5 varicose veins / CVI Symptomatic primary GSV, SSV or AASV incompetence, with reflux >0.5 seconds on colour duplex, including one or more of the following symptoms: aching, throbbing, heaviness,fatigue, pruritus, night cramps, restlessness, generalized pain or discomfort, swelling.

Patients who has GSV, SSV AASV diameters of 3mm to 12mm in the standing postition.

Only one limb of each patient was included in the study.

Exclusion Criteria:

- Current DVT or history of DVT. Recurrent varicose veins. Pregnant patients. Arterial disease (ABPI <0.8). Patients who are unwilling to participate this test. Inability or unwillingness to complete questionnaires. Adverse reaction to sclerosant or cyanoacrylate. GSV, SSV or AASV severely tortuous. Infectious disease. Life expectancy < 1 year. Current, regular use of systemic anticoagulation (e.g. warfarin, heparin). Daily use of narcotic analgesia or NSAIDS to control pain associated with venous disease.

The investigators determined that intravenous therapy was not appropriate.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-02-04 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-05 (Estimated)

PRIMARY OUTCOMES:
Technical Success at time of procedure | Immediately post-procedure
  Use duplex ultrasound assess the occlusion of treated vein post-procedure,record the rate of occlusion of treated vein post-procedure
Anatomical Success | 3days
  Use duplex ultrasound verify the occlusion of treated vessel and record the rate of occlusion of treated vessel
Anatomical Success | 12 months post-procedure
  Use duplex ultrasound verify the occlusion of treated vessel and record the rate of occlusion of treated vessel

SECONDARY OUTCOMES:
Instrumental success | Immediately post-procedure
  successful delivery of endovenous microwave ablation catheter in right place and successful withdrawal after microwave treatment is defined as Instrumental success
Quality of Life score using EQ-5D questionnaire | Baseline, 1 month, 6 months and 12 months
  EQ-5D is used to assess quality of life based on Mobility, Self-care, Usual Activities, Pain/Discomfort and Anxiety, rated at 5 levels: no problems, slight problems, moderate problems, severe problems, unable to perform activity. Inputs from this questionnaire is used to observe the changes in quality of life over the whole test procedure
Quality of life score using the Chronic Venous Insufficiency Questionnaire(CIVIQ-14) | Baseline, 1 month, 6 months and 12 months
  CIVIQ-14 is a questionnaire based on three dimensions - pain, physical and psychological, based on a scale from 1 to 5 (no trouble, slight, moderate, considerable, severe).Based on inputs, CIVIQ-14 will be tabulated, ranging from 0 to 100 - the higher the value, the poorer the quality of life.In order to observe the changes in quality of life over the whole test procedure.
Quality of life score using the Aberdeen Varicose Veins Questionnaire (AVVQ) | Baseline, 1 month, 6 months and 12 months
  To measure health status of varicose vein participants based on symptoms and impact on daily activities. A total score ranging from 0 to 30 will be tabulated, with 30 being worst quality of life.In order to observe the changes in quality of life over the whole test procedure.
Clinical Change using Venous Clinical Severity Score (VCSS) | Baseline, 1 month, 6 months and 12 months
  VCSS evaluates the severity of hallmarks of venous disease - 0 (none), 1 (Mild) , 2(Moderate), 3 (Severe).Record the score separately to observe the changes in quality of life over the whole test procedure.
Time taken to return to work and normal activities | 10 days post-op
  Investigators will make a call to follow up the day when the participants return to work and normal activities
Participants' satisfaction post-procedure | 3 days post-op
  To rate satisfaction with overall teatment regime with a numerical scale of 0 (least satisfied) to 10 (most satisfied) through an app named Recovery+

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of Chengdu University of Traditional Chinese Medicine, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gloviczki P, Comerota AJ, Dalsing MC, Eklof BG, Gillespie DL, Gloviczki ML, Lohr JM, McLafferty RB, Meissner MH, Murad MH, Padberg FT, Pappas PJ, Passman MA, Raffetto JD, Vasquez MA, Wakefield TW; Society for Vascular Surgery; American Venous Forum. The care of patients with varicose veins and associated chronic venous diseases: clinical practice guidelines of the Society for Vascular Surgery and the American Venous Forum. J Vasc Surg. 2011 May;53(5 Suppl):2S-48S. doi: 10.1016/j.jvs.2011.01.079. PMID 21536172
- [Result] Yang L, Wang X, Wei Z, Zhu C, Liu J, Han Y. The clinical outcomes of endovenous microwave and laser ablation for varicose veins: A prospective study. Surgery. 2020 Nov;168(5):909-914. doi: 10.1016/j.surg.2020.06.035. Epub 2020 Aug 10. PMID 32792099
- [Result] Yang L, Wang XP, Su WJ, Zhang Y, Wang Y. Randomized clinical trial of endovenous microwave ablation combined with high ligation versus conventional surgery for varicose veins. Eur J Vasc Endovasc Surg. 2013 Oct;46(4):473-9. doi: 10.1016/j.ejvs.2013.07.004. Epub 2013 Aug 1. PMID 23911734
- [Result] Liu D, Brace CL. Evaluation of tissue deformation during radiofrequency and microwave ablation procedures: Influence of output energy delivery. Med Phys. 2019 Sep;46(9):4127-4134. doi: 10.1002/mp.13688. Epub 2019 Jul 17. PMID 31260115
- [Result] Brace CL. Microwave ablation technology: what every user should know. Curr Probl Diagn Radiol. 2009 Mar-Apr;38(2):61-7. doi: 10.1067/j.cpradiol.2007.08.011. PMID 19179193
- [Result] Proebstle TM, Vago B, Alm J, Gockeritz O, Lebard C, Pichot O. Treatment of the incompetent great saphenous vein by endovenous radiofrequency powered segmental thermal ablation: first clinical experience. J Vasc Surg. 2008 Jan;47(1):151-156. doi: 10.1016/j.jvs.2007.08.056. PMID 18178468
- [Result] Quehe P, Alavi Z, Kurylo-Touz T, Saliou AH, Badra A, Baudino L, Gladu G, Ledan F, Haudebourg R, Gestin S, Bressollette L. Endovenous Celon radiofrequency-induced thermal therapy of great saphenous vein: A retrospective study with a 3-year follow-up. SAGE Open Med. 2018 Aug 21;6:2050312118794591. doi: 10.1177/2050312118794591. eCollection 2018. PMID 30891243
- [Result] Lawson JA, Gauw SA, van Vlijmen CJ, Pronk P, Gaastra MTW, Tangelder MJ, Mooij MC. Prospective comparative cohort study evaluating incompetent great saphenous vein closure using radiofrequency-powered segmental ablation or 1470-nm endovenous laser ablation with radial-tip fibers (Varico 2 study). J Vasc Surg Venous Lymphat Disord. 2018 Jan;6(1):31-40. doi: 10.1016/j.jvsv.2017.06.016. Epub 2017 Aug 24. PMID 29248107
- [Result] Simon CJ, Dupuy DE, Mayo-Smith WW. Microwave ablation: principles and applications. Radiographics. 2005 Oct;25 Suppl 1:S69-83. doi: 10.1148/rg.25si055501. PMID 16227498
- [Result] Vogl TJ, Naguib NN, Lehnert T, Nour-Eldin NE. Radiofrequency, microwave and laser ablation of pulmonary neoplasms: clinical studies and technical considerations--review article. Eur J Radiol. 2011 Feb;77(2):346-57. doi: 10.1016/j.ejrad.2009.07.034. Epub 2009 Aug 22. PMID 19700254
- [Derived] Zhang L, Lin Y, Geng C, Huang W, Yang Q, He C, Zeng W. Safety and efficacy of endovenous microwave ablation for treatment of varicose veins of the lower limbs in China: A prospective registered clinical trial. Vascular. 2025 Oct;33(5):1011-1019. doi: 10.1177/17085381241273225. Epub 2024 Aug 26. PMID 39183572